CLINICAL TRIAL: NCT06127940
Title: K-SAB Trial - Sotorasib Followed by SBRT to 1-3 Lesions in Advanced NSCLC With KRASG12C Mutation
Acronym: K-SAB
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: Sahlgrenska University Hospital (Other); Amgen (Industry)
Responsible Party: Principal Investigator, Karin Lindberg, Principal investigator, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K-SAB
Record Dates: First submitted 2023-10-04; First posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Non-small Cell Lung Cancer Metastatic
Keywords: Stereotactic body radiation therapy; KRAS-G12C mutation; NSCLC
MeSH Terms: interventions — Radiosurgery; sotorasib; GC Temporary Stopping

STUDY DESIGN:
Intervention Model Description: Single arm phase I study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Radiotherapy + sotorasib (Experimental): Sotorasib is administered as an 8-week-introduction treatment and if response on a CT-scan is observed (stable disease or partial response), the patient is treated with stereotactic radiation therapy (SBRT) to 1-3 of the remaining lesions.
  Interventions: Radiation: Stereotactic body radiation therapy (SBRT); Drug: Temporary Stopping

INTERVENTIONS:
Radiation: Stereotactic body radiation therapy (SBRT) — SBRT is delivered using institutional standard dosing while sotorasib is withheld during radiation.
  Other Names: Sotorasib
Drug: Temporary Stopping — Temporary stop of sotorasib during SBRT

SUMMARY:
The goal of this interventional study is to learn about the combination of sotorasib and stereotactic radiation therapy (SBRT) in patients with metastatic non-small cell lung cancer (NSCLC) with KRASG12C mutations. The main question it aims to answer is:

• can SBRT be safely delivered in patients treated with sotorasib

Participants will be treated with sotorasib for an 8-week-induction period and if the patient has stable disease or partial response, 1-3 of the remaining lesions will be irradiated with SBRT and sotorasib will then be contiuned after irradiation. The patients will then be followed and evaluated for toxicity to identify if grade 3-5 toxicity attributed to SBRT occurs within 6 months post SBRT. Tumour effects measured according to RECIST v1.1 will also be evaluated.

DETAILED DESCRIPTION:
Eligible subjects are those with a diagnosis of advanced KRASG12C mutated NSCLC who have received at least one line of standard medical treatment with immuno(chemo)therapy.

The subjects start with sotorasib and in parallel, 2-5 target lesions which are technically feasible to treat with SBRT, are identified. After 8 weeks of induction treatment of with sotorasib, the subjects are radiologically evaluated and subjects with stable disease (SD) or partial response (PR) on sotorasib will receive SBRT to minimum 1 and maximum 3 of the predefined lesions. Sotorasib is withheld during SBRT and then restarted after SBRT.

Sotorasib will continue until progression or other discontinuation criteria are met. The patients are followed clinically every month during the first 6 months post SBRT and then every 2-3 months. Radiological evaluation is performed every 2 months during the first year.

After the first 10 treated patients, a safety review meeting will be held and a decision whether to include 10 more patients will be performed.

ELIGIBILITY:
Main inclusion criteria:

1. Histological or cytological confirmed advanced NSCLC
2. KRASG12C mutation
3. Previous at least one line of treatment with immune- or/and chemotherapy or contraindications for immune- and/or chemotherapy.
4. Adequate organ function to tolerate sotorasib (see section 6.1 and 6.2 for details)
5. 2-5 lesions technically amenable to SBRT with 15 Gy x 3, 10 Gy x 5, or 7-8 Gy x 5.
6. Adequate organ function to tolerate SBRT:

   o Fulfilment of dose constraints to adequate organs at risk
7. ECOG performance status (PS) 0-1
8. FEV1 ≥1 litre (only applicable for lung targets)
9. Age ≥ 18 years
10. Measurable lesions according to RECIST

Main exclusion criteria:

1. Leptomeningeal carcinosis (on MRI or in cerebrospinal fluid) or metastases in the central nervous system
2. Previous RT for any cancer within the last 3 years possibly interfering with the planned RT within this study
3. Life expectancy of less than 6 months
4. Inability to understand given information or undergo study procedures according to protocol
5. Has evidence or a past medical history of interstitial lung disease or active, non-infectious pneumonitis or known pulmonary fibrosis
6. Woman who is pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 7 days after the last dose of sotorasib
7. Women of childbearing potential (WOCBP) unwilling to use a highly effective method of contraception during treatment and for an additional 7 days after the last dose of sotorasib. WOCBP using hormonal contraceptives should also use a barrier method
8. WOCBP with a positive pregnancy test assessed at screening or day 1 by a serum pregnancy test and/or urine pregnancy test
9. Centrally located pulmonary target (i.e., within 1 cm of the main bronchi or intermedius bronchus) and targets located within 1 cm of the gut, for SBRT
10. Use of known cytochrome P450 (CYP) 3A4 or P-gp sensitive substrates (with a narrow therapeutic window), within 14 days or 5 half-lives of the drug or its major active metabolite, whichever is longer, prior to study day 1 that was not reviewed and approved by the principal investigator
11. Use of strong inducers of CYP3A4 (including herbal supplements such as St. John´s wort) within 14 days or 5 half-lives, whichever is longer, prior to study day 1 that was not reviewed and approved by the principal investigator
12. Use of proton pump inhibitors (PPIs) within 3 days or H2-receptor antagonists within 1 day prior to study intervention
13. Use of warfarin. Use of Direct-Acting Oral Anticoagulants (DOAC) within 14 days or 5 half-lives, whichever is longer, prior to study day 1. Other anticoagulation may be allowed with principal investigator approval.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Safety - Grade 3 - 5 toxicity attributed to SBRT | 6 months post SBRT
  The number of patients presenting with grade 3-5 toxicity (attributed to SBRT) within 6 months post SBRT.

SECONDARY OUTCOMES:
Progression free survival | 1 year
  The number of patients who have progressed or died during the first 12 months post start of sotorasib (estimated using the KM-method).
Duration of response | 1 year
  The time between the date of first observation of CR or PR and the date of documented progressive disease for evaluable subjects. In all other situations, observations will be censored, or analysis only performed on those subjects who achieve a response.
Overall survival | 1 year
  The number of patients who have died during the first 12 months post start of sotorasib (estimated using the KM-method).
Overall toxicity related to SBRT | 1 year
  No and percentage of patients suffering toxicity attributed to SBRT (early toxic effects presenting within 3 months of finalization of SBRT vs late toxic effects presenting after more than 3 months post completion of SBRT).
Overall toxicity related to sotorasib | 1 year
  No and percentage of patients suffering toxicity attributed to sotorasib (early toxic effects presenting within 3 months of finalization of SBRT vs late toxic effects presenting after more than 3 months post completion of SBRT).

OTHER OUTCOMES:
Exploratory outcome | 1 year
  Prevalence of intrinsic and induced resistance mechanisms in response to KRASG12C inhibition with sotorasib.

CONTACTS AND LOCATIONS:
Overall Officials: Karin Lindberg, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Solna, Sweden